CLINICAL TRIAL: NCT01983358
Title: A Phase I Clinical Study, Randomized, Double-blind, Placebo-controlled,Single Dose, Dose Escalation Study of the Safety, Tolerability and Pharmacokinetics of JPI-289 in Healthy Male Subjects.
Brief Title: The Evaluation of Safety, Tolerability and Pharmacokinetics of Stroke Targeting Drug in Healthy Volunteers
Acronym: JPI-289
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: JP-NC-P1-13
Record Dates: First submitted 2013-11-04; First posted 2013-11-14 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2014-09

CONDITIONS: Stroke
Keywords: PARP-1 inhibitor
MeSH Terms: conditions — Stroke | interventions — JPI-289

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- JPI-289 (Experimental): Each cohort, volunteers will be infused JPI-289 through I.V for 30 min.(6 volunteers per each cohort, total 7 cohort)
  Interventions: Drug: JPI-289
- Placebo (Placebo Comparator): Each cohort, volunteer will be infused placebo through I.V for 30 min.(2 volunteers per each cohort, total 7 cohort)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: JPI-289 — PARP-1 inhibitor
  Arms: JPI-289
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study in to evaluate safety, tolerability, pharmacokinetics of JPI-289 in healthy male subjects.

DETAILED DESCRIPTION:
tPA treatment should be used within 3 hours after stroke onset for treating efficacy, but JPI-289 treatment(PARP-1 inhibitor) showed treating efficacy more than 10 hours after stroke onset. PARP-1 inhibitor add-on therapy of tPA will be very useful to prevent social, economic loss from physical, and mental disable by stroke.

This clinical trial progresses to explore safety, tolerability, pharmacokinetic/pharmacodynamic properties of JPI-289 by single dose escalation(7cohort). Investigational product medication of each level within 4 weeks evaluate safety and tolerability of patient through Data Safety Monitoring Board(DSMB) which is composed of more than 3 experts except principal investigator until the last visit. In each level 6 patients for investigational product and 2 patients for placebo will be allocated respectively in double blind manner.

ELIGIBILITY:
Inclusion Criteria:

* 19~55 years healthy male
* BMI measurement 20kg/m²~27kg/m²
* 90 ≤ SBP<140(mmHg) 60 ≤ DBP<100(mmHg) 45 ≤ Pulse rate<100(bpm)
* Signed the informed consent from to participate voluntarily and to comply with the trial requirements
* For a follow-up visit and during the study period, blood samples and availability

Exclusion Criteria:

* History of clinically significant hepatic, gastrointestinal, pulmonary, musculoskeletal, endocrine, psychiatric, hematooncologic, cardiovascular (Specially asthma, obstructive pulmonary disease, peptic ulcer)
* History of skin disease of graft affecting absorption of the drug
* History of drug abuse
* Positive urine drug screening
* Administrated investigational product in a previous clinical trial within 60 days of the screening test
* Donated blood within 60 days prior to screening test

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Difference of ECG, vital sign and diagnostic test in JPI-289 group and placebo group | -21d~9d

SECONDARY OUTCOMES:
Difference of concentration of JPI-289 in Plasma between JPI-289 group and placebo group | 0h~48h , 15 points
  * Blood
  * Urine 0h(pre-dose), 5min, 10min, 20min, 30min(before termination of infusion JPI-289), 45min, 1h, 2h, 4h, 8h, 12h, 24h, 48h

OTHER OUTCOMES:
Difference of PAR level in PBMC between JPI-289 group and placebo group | 0h(pre-dose)~48h, 6 points
  -Blood 0h(pre-dose),1h, 4h, 7h, 24h, 48h

CONTACTS AND LOCATIONS:
Overall Officials: HyeongSeok Lim, M.D.,Ph.D., Principal Investigator — AIDS Malignancy Consortium
Locations (1):
- Asan Medical Center, Seoul, Song-Pa Gu, South Korea

IPD SHARING:
Plan to Share IPD: No